CLINICAL TRIAL: NCT01852786
Title: Metabolic, Androgen, Blood Coagulation Parameters and Female Sexual Function in Relation to Oral Contraceptive Use and Androgen Receptor Polymorphisms in Healthy Lithuanian Women
Brief Title: The Effect of Hormonal Contraception on Female
Acronym: HORMCONTRA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Lithuanian University of Health Sciences (Other)
Responsible Party: Principal Investigator, Lina Ciaplinskiene, PhD student, Lithuanian University of Health Sciences
Other Study IDs: Contraception; contraception2013 (Registry Identifier: Lina Ciaplinskiene)
Record Dates: First submitted 2013-04-29; First posted 2013-05-14 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Adverse Effect of Oral Contraceptives, Initial Encounter
Keywords: Contraception; Hyperandrogenism; Female sexual function
MeSH Terms: conditions — Hyperandrogenism | interventions — Contraceptives, Oral, Combined; Natural Family Planning Methods

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Lipidogram, glycemia;
  2. Hormonal analyses by radioimmunoassay method ׃ total testosterone (T), free testosterone (FT), sex hormone binding globulin (SHBG), dehidroepiandrosterone sulphate (DHEAs), thyrotropin hormone (TSH), free thyroxine (FT4);
  3. Blood coagulation test׃ clotting time according to Ovren, fibrinogen, aPTT.
  4. Total blood picture test;
  5. Androgen receptor (AR) polymorphism test.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Contraceptives, Oral, Combined: The women, presenting for hormonal contraception use and with no contraindications for hormonal therapy.
  Interventions: Other: Contraceptives, Oral, Combined
- Controls: The women, presenting for non- hormonal contraception- barrier contraception methods -BCM- or natural family planning methods- NFPM.
  Interventions: Other: Controls

INTERVENTIONS:
Other: Contraceptives, Oral, Combined — • The women, presenting for hormonal contraception use and with no contraindications for hormonal therapy, one of the two medicines registered in Lithuania will be administered׃ Daylette (20 micrograms of Ethinylestradiol and 3 mg of Drospirenone) or Lindynette (20 micrograms of Ethinylestradiol and 75 micrograms of Gestoden).
  Other Names: COMBINED ORAL CONTRACEPTIVES
  Groups: Contraceptives, Oral, Combined
Other: Controls — The women, The women presenting for non-hormonal contraception use, will be recommended BCM or NFPM.
  Other Names: NATURAL FAMILY PLANNING
  Groups: Controls

SUMMARY:
The aim- To evaluate the impact of combined oral contraceptives on women's psychosexual, metabolic, blood coagulation, hormonal and genetic measures.

Combined oral contraceptives (COCs) is still the most popular contraception method. It is possible to find a number of publications about their non-contraceptive benefits, also about their adverse events. Most researches are conducted during clinical trials, which are commissioned by pharmaceutical companies, in order to compare COCs of different composition. This study set out to assess the role of psychosexual, metabolic, endocrine, hormonal and genetic measures of low dose combined oral contraceptive users- 20 micrograms of Ethinylestradiol/3 mg of Drospirenone and 20 micrograms of Ethinylestradiol/75 micrograms of Gestoden. Because this study is not commercial, it is expected to obtain valuable objective data - there are very few comparative studies about the impact of COCs to woman's organism.

DETAILED DESCRIPTION:
The aim

To evaluate the impact of combined oral contraceptives on women's psychosexual, metabolic, blood coagulation, hormonal and genetic measures.

The objectives

1. To asses the relation of AR polymorphisms to metabolic, androgen, blood coagulation parameters and sexual function in hormonal contraceptive users.
2. To compare the changes of metabolic, coagulation and endocrine parameters between hormonal and non-hormonal contraceptive users.
3. To assess the impact of COCs on the quality of woman's sexual life and her psychological state.
4. To assess the correlation between sex hormones and women's metabolic, endocrine, psychological, sexual function.
5. To evaluate the influence of COCs on the blood coagulation parameters.
6. To determine the importance of androgen parameters in diagnosis of hyperandrogenism.

Materials and Methods Setting׃ The study will be conducted in Lithuanian University of Health Sciences during the period from 2013 to 2016 years.

4 visits will be proceeded during the study: the screening visit and 3 additional visits - an inclusion in the study visit, a visit after 3 months and a visit after 6 months.

The screening visit (0 visit)

During the screening visit women will be questioned during the routine life and medical history. They will undergo a routine general clinical and gynecological examination:

1. height/weight (for BMI calculation) and hip/waist measurements;
2. blood pressure (BP) measurement ant a cardiac auscultation (for heart rate (HR) testing);
3. auscultation of lungs and palpation of the abdomen;
4. assessment of possible veins varicose in the legs;
5. bimanual gynecological examination;
6. breasts palpation;
7. genital ultrasound examination to assess possible anatomical anomalies;
8. thyroid ultrasound examination. Women meeting the assessment criteria will be introduced with The Informed Consent Form. Women who signed The Informed Consent Form will be invited to come for the 1 visit.

   1. visit

Women will repeatedly undergo a routine general examination (BP, HR). Genital and thyroid ultrasound will be performed.

Visual methods to determine the degree of hirsutism, as originally described by Ferriman and Gallwey (F-G), will be performed. The density of terminal hairs at 9 different body sites will be scored from 0 to 4, and total score will be calculated. In addition to the F-G scoring, the height/weight & hip/waist measurements, will be recorded. Hirsutism will be diagnosed in case of F-G≥8 scores.

* The women, presenting for hormonal contraception use and with no contraindications for hormonal therapy, one of the two medicines registered in Lithuania will be administered׃ Daylette (20 micrograms of Ethinylestradiol and 3 mg of Drospirenone) or Lindynette (20 micrograms of Ethinylestradiol and 75 micrograms of Gestoden).
* The women, presenting for non-hormonal contraception use, will be recommended barrier copntraception use(BCM),or Natural family planing methods (NFPM).

Women will be given to fill in six questionnaires׃

1. General questionnaire, developed by the authors to find out sociodemographic status;
2. Anxiety and Depression Scale (HAD)- to determine the level of anxiety and depression;
3. WHO-Five Wellbeing Index (WHO- 5)- to evaluate woman's well being;
4. Big Five- to assess personality traits;
5. Female Sexual Function Index (FSFI)- to find out the details of their sexual life;
6. Dyadic Adjustment Scale (DAD)- to assess the compatibility of the sexual partners.

Following blood tests will be performed׃

1. Lipogram, glycemia;
2. Hormonal analyses by radioimmunoassay method ׃ total testosterone (T), free testosterone (FT), sex hormone binding globulin (SHBG), dehydroepiandrosterone sulphate (DHEAs), thyrotropin hormone (TSH), free thyroxine (FT4);
3. Blood coagulation test׃ clotting time according to Ovran, fibrinogen,activated partial thromboplastin time (aPTT).
4. Total blood picture test;
5. Androgen receptor (AR) polymorphism test. Patients will be invited to come for another visit after 3 months. 2 visit

Women, arriving after 3 months, will be interwied about the changes in well-being and the potential side effects caused by the COCs. Women will undergo a routine general examination BP, HR, height/weight & hip/waist measurements). Genital and thyroid ultrasound will be performed. The signs of hyperandrogenism will be assessed using F-G scoring system.

Women will be given to fill in six questionnaires׃

1. Anxiety and Depression Scale;
2. WHO-Five Wellbeing Index;
3. Big Five;
4. Female Sexual Function Index;
5. Dyadic Adjustment Scale;
6. Satisfaction Questionnaire- to assess side effects, caused by used contraceptive method.

Patients will be invited to come for another visit after 6 months. 3 visit Women, arriving after 6 months, will be interwied about the changes in well-being and the potential side effects caused by the COCs. Women will undergo a routine general examination BP, HR, height/weight & hip/waist measurements). The signs of hyperandrogenism will be assessed using F-G scoring system.

Women will be given to fill in six questionnaires׃

1. Anxiety and Depression Scale;
2. WHO-Five Wellbeing Index;
3. Big Five;
4. Female Sexual Function Index;
5. Dyadic Adjustment Scale;
6. Satisfaction Questionnaire. Following blood tests will be performed׃

1. Lipogram, glycemia; 2. Hormonal analyses by radioimmunoassay method ׃ T, FT, SHBG, DHEAs, TSH, FT4; 3. Blood coagulation tests׃ clotting time according to Ovran, fibrinogen, aPTT; 4. Total blood picture test.

For further use of COCs patients will consult with the gynecologist performing the study.

ELIGIBILITY:
Inclusion Criteria:

1. 18 - 40 years old women applying to obstetrician-gynaecologist for contraception use or for preventive health care and giving their consent to participate in the study (who signed The Informed Consent Form) will be eligible to participate in the study. It is important to note that these women should not have underlying medical conditions (chronic non - infection diseases, chronic or acute infection diseases).
2. Not using hormonal contraception for 6 months or more.

Exclusion Criteria:

1. Women applying for obstetrician-gynaecologist consultation on gynaecological pathology.
2. Women with underlying medical conditions (chronic non - infection diseases, chronic or acute infection diseases).
3. Women, planning to get pregnant during the 12 months.
4. Pregnant women (suspected or confirmed pregnancy).

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 340 healthy Lithuanian women age 18- 40 years with regular menstruale cycle (22- 35 days) presenting for routine gynecologic concern or contraception purposes.
Sampling Method: Probability Sample
Enrollment: 340 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
Hirsutism | 2 years
  The expression of terminal hair growth using Ferriman- Gallwey scoring system in Lithuanian women will be assessed.

SECONDARY OUTCOMES:
Blood coagulation parameters and hormonal contraception | 3 years
  Blood coagulation parameters in six month period will be measured. The risk for development of thromboembolic complications for COCs use will be evaluated.
Lipids concentration | 3 years
  Changes of lipids concentration in COCs users will be identified.
Homeostasis model assessment | 3 years
  Having the results of the glucose concentration in the blood and fasting insulin level tests, the homeostasis model assessment (HOMA) will be calculated and evaluated dynamic changes of this measurement, while using COCs.
Free androgen Index | 3 years
  Having the results of the T and SHBG in the blood Free Androgen Index (FAI) will be calculated. We will compare the effectiveness of diagnostic methods, such as serum free testosterone measured by ELISA-method and free androgen index for assessment of hyperandrogenism in young women with hirsutism.

OTHER OUTCOMES:
Sexual function and hormonal contraception | 3 years
  The investigation should give answers to the questions of female sexual behavior, the quality of their sexual life and about the influence of COCs on the female mood and sexuality. The female sexual function and its disorders have not been investigated in Lithuania for young female group. The data of such investigation could become the basis for the sexual help centre and the diagnostics would improve.
Androgen receptor polymorphism and hormonal contraception | 3 years
  The relationship of androgen receptor - AR- repeat length in the AR gene will be evaluated.
AR gene polymorphism and metabolic function. | 3 yeras
  The correlation between AR gene polymorphism on metabolic function will be assessed.
AR gene polymorphism and endocrine function | 3 years
  The correlation between AR gene polymorphism on endocrine function will be assessed.
AR gene polymorphism and blood coagulation parameters | 3 years
  The correlation between AR gene polymorphism on blood coagulation parameters will be assessed.
AR gene polymorphism and psychosexual function | 3 years
  The correlation between AR gene polymorphism on psychosexual function will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Birute Zilaitiene, Ass. Proff., Principal Investigator — Lithuanian University of Health Sciences, Institute of Endocrinology
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania